CLINICAL TRIAL: NCT01701154
Title: The Effects of Respiratory Muscle Strength Training (RMST) on Inspiratory and Expiratory Muscle Strength in Adults and Children With Pompe Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00024468
Record Dates: First submitted 2012-10-03; First posted 2012-10-04 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Pompe Disease
Keywords: Pompe respiratory
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pompe: Adults and children with Pompe disease.
  Interventions: Other: respiratory muscle strength training

INTERVENTIONS:
Other: respiratory muscle strength training

SUMMARY:
The purpose of the study is to determine if respiratory muscle strength training will be beneficial for inspiratory and expiratory muscle strength in adults and children with Pompe disease.

DETAILED DESCRIPTION:
Respiratory muscle weakness results in substantial morbidity and mortality in individuals with almost all forms of neuromuscular disease (NMD), including both the infantile and adult phenotypes of Pompe disease. Although individual patterns of involvement vary, respiratory weakness in Pompe disease typically affects both the inspiratory and expiratory muscle systems. Our pilot data in two individuals with late-onset Pompe disease suggest that RMST may be a treatment for the progressive respiratory weakness encountered in this condition.

Purpose of the Study

* Determine the effect of respiratory muscle strength training on maximum inspiratory pressure, maximum expiratory pressure, upright % predicted forced vital capacity, and aspects of cough function.
* Determine the effect of RMST on functional outcome measures of gross motor function appropriate for individual participants in terms of age and motor skills.

ELIGIBILITY:
Inclusion Criteria:

* include skin fibroblast acid α-glucosidase (GAA) activity ≤1% of the normal mean, a minimum age of 3 years, the ability to participate in an intensive RMST research program, and the ability to maintain a consistent amount of nonresearch related physical activity over the course of the study.

Exclusion Criteria:

* include medical problems which preclude meaningful participation in the study, the inability to perform high effort respiratory tasks using maximum intensity, respiratory weakness so profound that RMST cannot be completed at the minimum pressure thresholds of available respiratory trainers, and the inability to safely perform the protocol. For example, high effort respiratory tasks are occasionally associated with mild, transient dizziness which quickly dissipates following a brief rest. If severe and/or prolonged dizziness were to occur in a particular case, then exclusion from the study would be necessary.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with Pompe disease
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12-15 (Actual); Study Completion 2012-12-15 (Actual)

PRIMARY OUTCOMES:
Change in maximum inspiratory pressure | baseline, week 12
  change from pre-test to post-test

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Jones, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States